CLINICAL TRIAL: NCT00454870
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-Center Study of the Pharmacodynamics/Efficacy, Safety, Tolerability, and Pharmacokinetics of 3 Fixed Dosages of MEM 3454 (5 mg, 15 mg, and 50 mg) in Patients With Mild to Moderate Alzheimer's Disease
Brief Title: Safety and Efficacy of MEM 3454 Versus Placebo in Patients With Mild to Moderate Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memory Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEM 3454-003
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Last update posted 2008-05-06 (Estimated); Status verified 2008-05

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; Cognition; Cognitive impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MEM 3454

SUMMARY:
The purpose of this study is to determine in an 8-week treatment study if MEM 3454 is a safe and effective treatment for patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
Alzheimer's disease is the leading cause of dementia and one of the most common diseases of the aging population. It is a chronic brain disease that involves gradual memory loss, decline in the ability to perform routine tasks, disorientation, difficulty in learning, loss of language skills, impairment of judgment, and personality changes in affected individuals. The neurodegenerative nature of the disease eventually leads to the failure of other organ systems and death.

A consistent and marked change in the brains of patients with AD is degeneration of the cholinergic innervation in the hippocampus and cerebral cortex areas. The activity of choline acetyl transferase (ChAT) is significantly reduced in these brain regions, and a linear correlation is seen between the reduction in cortical ChAT activity and the progress of dementia, indicating a progressive loss of cholinergic function.

Receptor selective nicotinic alpha-7 receptor agonists can modulate acetylcholine in selective brain regions and contribute to symptomatic treatment of AD. MEM 3454 is a novel nicotinic alpha-7 receptor selective partial agonist having serotonin type 3 (5-HT3) receptor antagonist properties.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or possible Alzheimer's disease
* MMSE score between 16 and 26 points
* Modified Hachinski Ischemia Score of less than or equal to 4
* Capable of performing cognitive tests and other procedures specified in protocol

Exclusion Criteria:

* Head trauma associated with cognitive impairment
* Evidence of significant neurological disease other than AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, CNS tumor, progressive supranuclear palsy, seizure disorder, etc.
* Received AChE inhibitor therapy (e.g., rivastigmine, tacrine or galantamine) or NDMA-receptor antagonist, memantine, within 30 days or donepezil within 40 days of randomization
* Received any investigational drug within 2 months of randomization or treatment with other nicotinic receptor agonists within 3 months of screening

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-02; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Murray, MD, PhD, Study Director — Memory Pharmaceuticals Corp
Locations (6):
- United States (6):
  - Phoenix, Arizona
  - Glendale, California
  - Atlanta, Georgia
  - Wichita, Kansas
  - Willingboro, New Jersey
  - Philadelphia, Pennsylvania